CLINICAL TRIAL: NCT02309125
Title: Split Mouth Clinical Study to Compare the Secondary Stability of Dental Implants Using Immediate Gradual Loading Versus Early Loading Protocol in Posterior Maxilla. A Randomized Controlled Trial
Brief Title: Comparing the Secondary Stability of Dental Implants: Immediate Gradual Loading Versus Early Loading Protocol in Posterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elhassan Mohamed Elsayed Mostafa Mossad, Master student, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: immediate_early_loading
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Dental Implant; Transmucosal Healing; Bone Loss
Keywords: immediate gradual loading
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- implant A (Experimental): will include implants with immediate progressive loading using gingival formers of different sizes
  Interventions: Procedure: immediate progressive loading using gingival formers
- implant B (Other): The implants will remain submerged from surgery time till loading time 2 month.(submerged healing)
  Interventions: Procedure: submerged healing

INTERVENTIONS:
Procedure: immediate progressive loading using gingival formers — Implant placement will be 1 mm subcrestally, and it will receive transmucosal healing using gingival former.
  The gingival former will be replaced every 2 weeks by consequent larger size gingival former (at surgery time group A will receive 2 mm height gingival former which will be swapped by,3 mm, 4 mm and the last is 5 mm).
  Arms: implant A
Procedure: submerged healing — the implant placement will be 1 mm subcrestally, and it will receive unloaded healing.(submerged healing)
  Arms: implant B

SUMMARY:
The aim of this split mouth study is to compare which method is better in reducing bone loss and healing times following implants. Specifically, the two methods investigated will be immediate gradual loading and early loading protocol.

Research Hypothesis Immediate gradual loading using gingival formers is superior to early loading protocols in improving bone quality and thus reducing the healing time.

DETAILED DESCRIPTION:
These two methods (gradual loading and early loading) will both be used in implants patients with the aim to compare which protocol leads to a better outcome for the patient.

A 'better outcome' is defined as the method, which leads to the least crestal bone loss, and the fastest healing time.

Immediate gradually loaded side: will include transmucosal healing of dental implants using gingival formers which will be replaced every 2 weeks by consequent larger size gingival former.i.e. at surgery time the implants will receive 2 mm height gingival former which will be swapped by 3 mm, 4 mm, 5 mm and the last is 6 mm

early loaded side: implants will be submerged from the surgery time till loading time (2 month).

ELIGIBILITY:
Inclusion criteria

1. Patients with bilateral Partial or complete edentulous areas in maxillary premolar/molar region.
2. Free medical history.
3. Enough bone quantity.
4. Enough keratinized mucosa

Exclusion criteria

1. Systemic disease.
2. Irradiated bone (radiotherapy).
3. Heavy smoking habit.
4. Patients undergoing long-term immunosuppressive therapy.
5. Atrophic ridges.
6. Presence of any local bony lesion.
7. Presence of mandibular parafunctional habits

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
secondary stability of dental implant (ISQ Osstell Mentol) | 2 month
  ISQ Osstell Mentol

SECONDARY OUTCOMES:
Bone loss using Periapical Radiographic (Long Cone Paralleling technique) | 2 month
  using Periapical Radiographic (Long Cone Paralleling technique)

CONTACTS AND LOCATIONS:
Overall Officials: elhassan mossad, oral surgeon, Principal Investigator — Cairo University
Locations (1):
- Faculty of oral & Dental Medicine. Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Appleton RS, Nummikoski PV, Pigno MA, Cronin RJ, Chung KH. A radiographic assessment of progressive loading on bone around single osseointegrated implants in the posterior maxilla. Clin Oral Implants Res. 2005 Apr;16(2):161-7. doi: 10.1111/j.1600-0501.2004.01089.x. PMID 15777325
- [Background] Attard NJ, Zarb GA. Immediate and early implant loading protocols: a literature review of clinical studies. J Prosthet Dent. 2005 Sep;94(3):242-58. doi: 10.1016/j.prosdent.2005.04.015. PMID 16126077
- [Background] Berglundh T, Abrahamsson I, Lindhe J. Bone reactions to longstanding functional load at implants: an experimental study in dogs. J Clin Periodontol. 2005 Sep;32(9):925-32. doi: 10.1111/j.1600-051X.2005.00747.x. PMID 16104954
- [Background] Buchter A, Wiechmann D, Koerdt S, Wiesmann HP, Piffko J, Meyer U. Load-related implant reaction of mini-implants used for orthodontic anchorage. Clin Oral Implants Res. 2005 Aug;16(4):473-9. doi: 10.1111/j.1600-0501.2005.01149.x. PMID 16117773
- [Background] Duyck J, Vandamme K, Geris L, Van Oosterwyck H, De Cooman M, Vandersloten J, Puers R, Naert I. The influence of micro-motion on the tissue differentiation around immediately loaded cylindrical turned titanium implants. Arch Oral Biol. 2006 Jan;51(1):1-9. doi: 10.1016/j.archoralbio.2005.04.003. Epub 2005 May 31. PMID 15922992
- [Background] Duyck J, Vrielinck L, Lambrichts I, Abe Y, Schepers S, Politis C, Naert I. Biologic response of immediately versus delayed loaded implants supporting ill-fitting prostheses: an animal study. Clin Implant Dent Relat Res. 2005;7(3):150-8. doi: 10.1111/j.1708-8208.2005.tb00059.x. PMID 16219245
- [Background] Ghoveizi R, Alikhasi M, Siadat MR, Siadat H, Sorouri M. A radiographic comparison of progressive and conventional loading on crestal bone loss and density in single dental implants: a randomized controlled trial study. J Dent (Tehran). 2013 Mar;10(2):155-63. Epub 2013 Mar 31. PMID 23724215
- [Background] Isidor F. Mobility assessment with the Periotest system in relation to histologic findings of oral implants. Int J Oral Maxillofac Implants. 1998 May-Jun;13(3):377-83. PMID 9638008
- [Background] Piattelli A, Corigliano M, Scarano A, Costigliola G, Paolantonio M. Immediate loading of titanium plasma-sprayed implants: an histologic analysis in monkeys. J Periodontol. 1998 Mar;69(3):321-7. doi: 10.1902/jop.1998.69.3.321. PMID 9579618
- [Background] Piattelli A, Scarano A, Piattelli M, Bertolai R, Panzoni E. Histologic aspects of the bone and soft tissues surrounding three titanium non-submerged plasma-sprayed implants retrieved at autopsy: a case report. J Periodontol. 1997 Jul;68(7):694-700. doi: 10.1902/jop.1997.68.7.694. PMID 9249642
- [Background] Soballe K, Hansen ES, Brockstedt-Rasmussen H, Hjortdal VE, Juhl GI, Pedersen CM, Hvid I, Bunger C. Gap healing enhanced by hydroxyapatite coating in dogs. Clin Orthop Relat Res. 1991 Nov;(272):300-7. PMID 1657476
- [Background] Szmukler-Moncler S, Piattelli A, Favero GA, Dubruille JH. Considerations preliminary to the application of early and immediate loading protocols in dental implantology. Clin Oral Implants Res. 2000 Feb;11(1):12-25. doi: 10.1034/j.1600-0501.2000.011001012.x. PMID 11168189
- [Background] Frost HM. Perspectives: bone's mechanical usage windows. Bone Miner. 1992 Dec;19(3):257-71. doi: 10.1016/0169-6009(92)90875-e. PMID 1472896
- [Background] Frost HM. A 2003 update of bone physiology and Wolff's Law for clinicians. Angle Orthod. 2004 Feb;74(1):3-15. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15038485
- [Background] Misch CE, Hoar J, Beck G, Hazen R, Misch CM. A bone quality-based implant system: a preliminary report of stage I & stage II. Implant Dent. 1998;7(1):35-42. doi: 10.1097/00008505-199804000-00004. PMID 9588972
- [Background] Jones HH, Priest JD, Hayes WC, Tichenor CC, Nagel DA. Humeral hypertrophy in response to exercise. J Bone Joint Surg Am. 1977 Mar;59(2):204-8. PMID 845205
- [Background] Martin B. Aging and strength of bone as a structural material. Calcif Tissue Int. 1993;53 Suppl 1:S34-9; discussion S39-40. doi: 10.1007/BF01673400. PMID 8275378
- [Background] Quinlan P, Nummikoski P, Schenk R, Cagna D, Mellonig J, Higginbottom F, Lang K, Buser D, Cochran D. Immediate and early loading of SLA ITI single-tooth implants: an in vivo study. Int J Oral Maxillofac Implants. 2005 May-Jun;20(3):360-70. PMID 15973947
- [Background] Roberts WE, Turley PK, Brezniak N, Fielder PJ. Implants: Bone physiology and metabolism. CDA J. 1987 Oct;15(10):54-61. No abstract available. PMID 3331974
- [Background] Degidi M, Iezzi G, Scarano A, Piattelli A. Immediately loaded titanium implant with a tissue-stabilizing/maintaining design ('beyond platform switch') retrieved from man after 4 weeks: a histological and histomorphometrical evaluation. A case report. Clin Oral Implants Res. 2008 Mar;19(3):276-82. doi: 10.1111/j.1600-0501.2007.01449.x. Epub 2007 Dec 13. PMID 18081870
- [Background] Diab T, Sit S, Kim D, Rho J, Vashishth D. Age-dependent fatigue behaviour of human cortical bone. Eur J Morphol. 2005 Feb-Apr;42(1-2):53-9. doi: 10.1080/09243860500095539. PMID 16123024